CLINICAL TRIAL: NCT03586271
Title: Comparison of the Visual Performance After Implantation of a Trifocal Intraocular Lens(AT Lisa Tri 839MP) and Two Bifocal Intraocular Lenses(ReSTOR +2.5/+ 3.0D and Diff-aay)
Brief Title: Comparison of the Visual Performance After Implantation of Multifocal Lens
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aier School of Ophthalmology, Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: SHIRB2018016
Record Dates: First submitted 2018-06-15; First posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-05

CONDITIONS: Intraocular Lens

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- trifocal lens: trifocal lens implantation(AT Lisa tri 839MP)
  Interventions: Procedure: bifocal lens 1; Procedure: bifocal lens 2; Procedure: bifocal lens 3
- bifocal lens 1: bifocal lens implantation(Diff-aay)
  Interventions: Procedure: trifocal lens; Procedure: bifocal lens 2; Procedure: bifocal lens 3
- bifocal lens 2: bifocal lens implantation(ReSTOR +3.0D)
  Interventions: Procedure: trifocal lens; Procedure: bifocal lens 1; Procedure: bifocal lens 3
- bifocal lens 3: bifocal lens implantation(ReSTOR +2.5D)
  Interventions: Procedure: trifocal lens; Procedure: bifocal lens 1; Procedure: bifocal lens 2

INTERVENTIONS:
Procedure: trifocal lens — phacoemusification + trifocal lens(AT Lisa tri 839MP) implantation
  Groups: bifocal lens 1; bifocal lens 2; bifocal lens 3
Procedure: bifocal lens 1 — phacoemusification +bifocal lens(Diff-aay) implantation
  Groups: bifocal lens 2; bifocal lens 3; trifocal lens
Procedure: bifocal lens 2 — phacoemusification +bifocal lens (ReSTOR +3.0D) implantation
  Groups: bifocal lens 1; bifocal lens 3; trifocal lens
Procedure: bifocal lens 3 — phacoemusification +bifocal lens (ReSTOR +2.5D) implantation
  Groups: bifocal lens 1; bifocal lens 2; trifocal lens

SUMMARY:
This is a prospective, consecutive, nonrandomized,comparative study. Comparison of the Visual Performance After Implantation of a Trifocal Intraocular Lens and Two Bifocal Intraocular Lenses

DETAILED DESCRIPTION:
Multifocal intraocular lenses were introduced in the 1980s and have the benefit of promoting near and far vision simultaneous. However, these multifocal lenses have the disadvantages, including lower contrast sensitivity(CS) and visual discomfort, such as halos, glares and starburst, et al. Therefore, careful patient selection is crucial to achieve good postoperative results. The purpose of this study was to compare the visual outcomes and subjective visual quality between bifocal intraocular Lens(ReSTOR +2.5/+ 3.0D and Diff-aay) and trifocal intraocular Lens(AT Lisa tri 839MP). This prospective, nonrandomized, consecutive, comparative study included the assessment of 60 patients implanted with multifocal intraocular lens. visual acuity was tested in all cases. Ophthalmological evaluation included the measurement of uncorrected distance visual acuity (UDVA), corrected distance visual acuity (CDVA), uncorrected near visual acuity (UNVA), and uncorrected intermediate visual acuity (UIVA), the analysis of contrast sensitivity (CS), visual defocus curve, spectacle independence, patient satisfaction, residual sphere, spherical equivalent (SE), cylinder and complications.

ELIGIBILITY:
Inclusion Criteria:

* cataract

Exclusion Criteria:

* existence of any corneal disease;
* previous eye surgery;
* illiteracy;
* previous refractive surgery;
* expected postoperative corneal astigmatism more than 1.00D;
* higer-order aberration more than 0.3;
* spherical aberration more than 0.3μm;
* intraoperative or postoperative complications.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cataract patients
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-08-02 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Uncorrected distance visual acuity | 3 months after surgery
  Uncorrected distance visual acuity (4m) were measured using the reading table model of the Early Treatment Diabetic Retinopathy Study charts (ETDRS; Vector Vision, Ltd, Greenville, OH, USA).
Uncorrected near visual acuity | 3 months after surgery
  Uncorrected near visual acuity (40cm) were measured using the reading table model of the Early Treatment Diabetic Retinopathy Study charts (ETDRS; Vector Vision, Ltd, Greenville, OH, USA).
Uncorrected intermediate visual acuity | 3 months after surgery
  Uncorrected intermediate visual acuity (60cm) were measured using the reading table model of the Early Treatment Diabetic Retinopathy Study charts (ETDRS; Vector Vision, Ltd, Greenville, OH, USA).

OTHER OUTCOMES:
Quality of vision | 3 months after surgery
  Quality of vision was measured using the National Eye Institute Visual Function Questionnaire (NEI VFQ)-25. The NEI-VFQ was developed at the RAND under the sponsorship of the NEI; it provides a self-reported measure of visual function.

CONTACTS AND LOCATIONS:
Overall Officials: Wensheng Li, Study Director — Shanghai Aier Eye Hosptial
Locations (1):
- Wensheng Li, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results
Supporting Information: Study Protocol, SAP
Time Frame: After this study is finished the data will become available for 1year.
Access Criteria: The analytical data will be accessed in published articles.

REFERENCES:
- [Background] de Medeiros AL, de Araujo Rolim AG, Motta AFP, Ventura BV, Vilar C, Chaves MAPD, Carricondo PC, Hida WT. Comparison of visual outcomes after bilateral implantation of a diffractive trifocal intraocular lens and blended implantation of an extended depth of focus intraocular lens with a diffractive bifocal intraocular lens. Clin Ophthalmol. 2017 Oct 26;11:1911-1916. doi: 10.2147/OPTH.S145945. eCollection 2017. PMID 29138533
- [Background] Gundersen KG, Potvin R. Comparison of visual outcomes after implantation of diffractive trifocal toric intraocular lens and a diffractive apodized bifocal toric intraocular lens. Clin Ophthalmol. 2016 Mar 17;10:455-61. doi: 10.2147/OPTH.S103375. eCollection 2016. PMID 27051269
- [Background] Xu Z, Cao D, Chen X, Wu S, Wang X, Wu Q. Comparison of clinical performance between trifocal and bifocal intraocular lenses: A meta-analysis. PLoS One. 2017 Oct 26;12(10):e0186522. doi: 10.1371/journal.pone.0186522. eCollection 2017. PMID 29073156